CLINICAL TRIAL: NCT02667704
Title: Influence of Bosentan on the Pharmacokinetics of Nintedanib in Healthy Male Subjects
Brief Title: Influence of Bosentan on the Pharmacokinetics of Nintedanib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1199.239; 2015-003819-38 (EudraCT Number: EudraCT)
Record Dates: First submitted 2016-01-21; First posted 2016-01-29 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Healthy
MeSH Terms: interventions — Bosentan; nintedanib

ARMS (2):
- Nintedanib (Experimental)
  Interventions: Drug: Nintedanib
- Bosentan (Experimental)
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan
  Arms: Bosentan
Drug: Nintedanib
  Arms: Nintedanib

SUMMARY:
The trial was designed to investigate whether, and to which extent, multiple doses of bosentan may influence the plasma levels of nintedanib administered as a single dose.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigators assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Males who are willing to use a medically acceptable method of contraception during the study (from start of treatment until end of trial examination). Acceptable methods of contraception for use by male volunteers include sexual abstinence, a vasectomy performed at least 1 year prior to dosing, and barrier contraception (condom). Subjects, who are not vasectomised or sexually abstinent have to ensure that an additional acceptable method of contraception will be used by his female partner such as IUD (intrauterine device), surgical sterilisation (including hysterectomy), hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first nintedanib administration, or barrier method (e.g. diaphragm with spermicide).

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Laboratory parameters ALT, AST or GGT outside the reference range
* Intake of drugs that inhibit the efflux of bile salts (e.g. rifampicin, glibenclamide, cyclosporine) within 30 days prior to administration of trial medication

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is open-label, mono-center clinical trial in healthy male subjects applied a fixed sequence, two-treatment, two- period crossover design. All subjects were to undergo 2 trial periods in a fixed sequence, receiving reference treatment (R) in Period 1, and test treatment (T) in Period 2. A wash-out between Periods 1 and 2 was not mandatory.
Groups:
- Nintedanib (Reference (R)) / Bosentan+Nintedanib (Test (T)): Subject received single dose of 150 milligram (mg) Nintedanib (1 x 1 soft gelatin capsule) on day 1 of period 1 and then multiple doses of 250 mg Bosentan (2 x 1 film-coated tablets) on days 1 to 8 of period 2 plus single dose of 150 milligram (mg) Nintedanib (1 x 1 soft gelatin capsule) on day 7 of period 2 administered orally with 240 millilitre (mL) of water
Period: Treatment Period 1
Arm/Group | Nintedanib (Reference (R)) / Bosentan+Nintedanib (Test (T))
Started | 13
Completed | 13
Not Completed | 0
Period: Treatment Period 2
Arm/Group | Nintedanib (Reference (R)) / Bosentan+Nintedanib (Test (T))
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS), full analysis set in the sense of ICH-E9: all subjects from the entered set (all subjects who entered the trial, whether treated or not) who were documented to have received 1 dose of trial medication.
Arm/Group | Nintedanib (Reference (R)) / Bosentan+Nintedanib (Test (T))
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.0 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Nintedanib in Plasma Over the Time Interval From 0 to the Last Quantifiable Concentration (AUC0-tz)
Description: Area under the concentration-time curve of Nintedanib in plasma over the time interval from 0 to the last quantifiable concentration (AUC0-tz). PK plasma samples were taken at: 1 hour (h) before drug administration (approximate time for predose sample) and 30 minutes, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h, 144h, 144.5h, 145h, 145.5h, 146h, 146.5h, 147h, 148h, 149h, 150h, 152h, 154h, 156h, 168h, 180h, 192h, 216h after drug administration. Two different visits; Visit 2 (R): -1 to 72 h, Visit 3 (T) 144 to 216 h. AUC0-tz was calculated for each visit separately.
Time Frame: Up to 216 hours. The details are mentioned in description.
Population: Pharmacokinetic parameter analysis set (PKS): all subjects in the treated set who provided at least one primary or secondary pharmacokinetic (PK) parameter not flagged for exclusion due to a protocol violation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)*hour (h) /millilitre (mL)
Groups:
- Nintedanib (R): Subject received single dose of 150 milligram (mg) Nintedanib (1 x 1 soft gelatin capsule) on day 1 administered orally with 240 millilitre (mL) of water.
- Bosentan+Nintedanib (T): Subject received multiple doses of 250 mg Bosentan (2 x 1 film-coated tablets) on days 1 to 8 plus single dose of 150 milligram (mg) Nintedanib (1 x 1 soft gelatin capsule) on day 7 administered orally with 240 mL of water
Arm/Group | Nintedanib (R) | Bosentan+Nintedanib (T)
Number analyzed (Participants) | 13 | 13
nanogram (ng)*hour (h) /millilitre (mL) | 195 (38.8) | 193 (33.4)
Statistical Analysis 1: Comparison: Nintedanib (R) vs Bosentan+Nintedanib (T); Analysis of variance (ANOVA) model on the log scale including treatment as fixed effect and subject as a random effect; Test type: Superiority or Other; ANOVA; Ratio of geometric means in percentage = 98.85, 90% CI 2-sided [91.320 to 107.010], Standard Deviation 11.4 — Relative bioavailability was estimated by the ratio (T/R) of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient of variation

2. Primary Outcome: Maximum Measured Concentration of Nintedanib in Plasma (Cmax)
Description: Maximum measured concentration of Nintedanib in plasma (Cmax). PK plasma samples were taken at: 1 hour (h) before drug administration and 30 minutes, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h, 144h, 144.5h, 145h, 145.5h, 146h, 146.5h, 147h, 148h, 149h, 150h, 152h, 154h, 156h, 168h, 180h, 192h, 216h after drug administration. Two different visits; Visit 2 (R): -1 to 72 h, Visit 3 (T) 144 to 216 h. Cmax was determined for each visit separately.
Time Frame: Up to 216 hours. The details are mentioned in description.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nintedanib (R) | Bosentan+Nintedanib (T)
Number analyzed (Participants) | 13 | 13
ng/mL | 21.9 (55.2) | 22.7 (42.2)
Statistical Analysis 1: Comparison: Nintedanib (R) vs Bosentan+Nintedanib (T); Analysis of variance (ANOVA) model on the log scale including treatment as fixed effect and subject as a random effect; Test type: Superiority or Other; ANOVA; Ratio of geometric means in percentage = 103.36, 90% CI 2-sided [86.134 to 124.025], Standard Deviation 26.5 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Concentration-time Curve of Nintedanib in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity)
Description: Area under the concentration-time curve of Nintedanib in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity). PK plasma samples were taken at: 1 hour (h) before drug administration and 30 minutes, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h, 144h, 144.5h, 145h, 145.5h, 146h, 146.5h, 147h, 148h, 149h, 150h, 152h, 154h, 156h, 168h, 180h, 192h, 216h after drug administration. Two different visits; Visit 2 (R): -1 to 72 h, Visit 3 (T) 144 to 216 h. AUC0-infinity was calculated for each visit separately.
Time Frame: Up to 216 hours. The details are mentioned in description.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h / mL
Arm/Group | Nintedanib (R) | Bosentan+Nintedanib (T)
Number analyzed (Participants) | 13 | 13
ng*h / mL | 204 (38.3) | 208 (34.1)
Statistical Analysis 1: Comparison: Nintedanib (R) vs Bosentan+Nintedanib (T); Analysis of variance (ANOVA) model on the log scale including treatment as fixed effect and subject as a random effect; Test type: Superiority or Other; ANOVA; Ratio of geometric means in percentage = 101.98, 90% CI 2-sided [94.909 to 109.570], Standard Deviation 10.3 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 13 days after the last drug administration, up to 21 days
Groups:
- Nintedanib (R): Subject received single dose of 150 milligram (mg) Nintedanib (1 x 1 soft gelatin capsule) on day 1 of period 1 administered orally with 240 millilitre (mL) of water.
- Bosentan: Subject received multiple doses of 250 mg Bosentan (2 x 1 film-coated tablets) on days 1 to 6 of period 2 administered orally with 240 mL of water
- Bosentan+Nintedanib (T): Subject received multiple doses of 250 mg Bosentan (2 x 1 film-coated tablets) on days 7 and 8 of period 2 plus single dose of 150 milligram (mg) Nintedanib (1 x 1 soft gelatin capsule) on day 7 administered orally with 240 mL of water
Arm/Group | Nintedanib (R) | Bosentan | Bosentan+Nintedanib (T)
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 4/13 | 4/13 | 2/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (R) (N=13) | Bosentan (N=13) | Bosentan+Nintedanib (T) (N=13)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: Other